CLINICAL TRIAL: NCT01502475
Title: A Survey of Complementary and Conventional Medicine Use Patterns in the Veteran Population
Acronym: CACMAS
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 11-1086
Record Dates: First submitted 2011-12-28; First posted 2011-12-30 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2012-07

CONDITIONS: Alternative Medicine; Attitudes; Beliefs; Veterans
Keywords: Complementary Alternative Medicine; Veteran; Attitudes; Beliefs
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Veteran Attitudes toward CAM

SUMMARY:
In this protocol, the investigators proposed to assess the Complementary Alternative Medicine (CAM) usage patterns in a Veteran population using a CAM survey developed by Dr. Hernandez and colleagues. This survey, the Complementary, Alternative and Conventional Medicines Attitudes Scale (CACMAS), is a brief, self-report questionnaire that assesses medical use patterns, as well as attitudes about medical treatment and the relationship among these. The CACMAS will assess the potential role of individual beliefs and attitudes towards complementary and conventional medicine usage patterns, and possibly indicate how this scale might be used to predict optimal treatment offerings for a particular population given attitudes about medical treatments.

DETAILED DESCRIPTION:
The use of complementary and alternative medicine (CAM) in the United States has seen a steady and steep rise over the past two decades. A national survey of over 31,000 adults found that 36% of respondents had used CAM therapies in the last month, and this estimate increased to 62% when prayer for health reasons was included. Second, this same survey showed that CAM is often used to treat symptoms and illnesses associated with stress such as depression, anxiety, back and neck pain, and gastrointestinal disorders. Finally, many individuals experiencing high levels of stress lack access to conventional medicine due to lack of medical insurance, possibly increasing the attractiveness of CAM for these individuals. This ongoing systematic characterization of CAM usage patterns in civilian populations has not been mirrored in active military and military Veteran populations across the United States. Data from the less than handful of studies that have been conducted thus far, suggest that CAM usage patterns in military and military Veteran populations are influenced by demographics and certain medical conditions, as well as dissatisfaction with certain aspects of conventional care. While there appears to be some similarity between civilian and non-civilians populations, there remains much to be known in the latter population.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18 and 89
* Currently eligible or receiving health care at a VA Medical Center

Exclusion Criteria:

* Inability to provide informed consent
* Inability to answer comprehension questions

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A range of Veterans eligible to, or seeking care, from a Veterans Affairs healthcare setting.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Conventional Medicine Attitudes Scale (CACMAS) | One time

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brenner, PhD, Principal Investigator — VA Eastern Colorado Health Care System
Locations (2):
- United States (2):
  - Denver Veterans Affairs Medical Center/VAECHCS, Denver, Colorado
  - Eastern Colorado Health Care System Denver VA, Denver, Colorado

REFERENCES:
- See also: Related Info — http://www.mirecc.va.gov/visn19/